CLINICAL TRIAL: NCT02054403
Title: Structural and Functional Parameters in Caucasian Patients With Angle Closure on SS-OCT
Brief Title: Angle Closure (Glaucoma) in Caucasians
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL47347.068.13/METC 13-2-060
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- angle closure

SUMMARY:
Rationale: Primary angle closure glaucoma (PACG) causes high rates of blindness, either by means of a painful attack of acute angle closure glaucoma or unnoticed over a period of many years. Patients with angle closure are particularly at risk but can be detected during an ophthalmological examination and sent for early preventive (laser) intervention. Current practice shows that patients at risk of PACG are frequently missed during routine examinations. Moreover, new imaging techniques like swept source optical coherence tomography (SS-OCT), are emerging with which the angle of the anterior chamber can be imaged in great detail with no burden for the patient. These techniques are already used in clinical practice and replace and complete part of the ophthalmic examination. However, in Caucasians, it is not yet known to what extent angle closure is detected in regular care and can be detected with this OCT device. There are few published data concerning angle closure and PACG in Caucasians and its characteristics.

Objective: To quantify the presence of angle closure by gonioscopy in patients at risk of angle closure on SS-OCT. Secondary objectives are to quantify the presence of an increased intra-ocular pressure during the day or after dark provocation, to quantify morphometric details of the anterior chamber, structural changes, and corneal endothelial cells and to quantify the functional changes of the visual field.

Study design: prospective, observational, descriptive study. Study population: Caucasian patients, presenting at the outpatient clinic of the University Eye Clinic Maastricht, aged 40 to 80 years, who are diagnosed with angle closure on SS-OCT.

Intervention (if applicable): Not applicable. Main study parameters/endpoints: The main study parameter is assessment of the anterior chamber angle according to gonioscopy. Secondary study parameters are the presence of an increased intra-ocular pressure (IOP) (>21 mmHg) during the day or after dark provocation (IOP rise from baseline), morphometric details of the anterior chamber, structural changes of the retinal nerve fiber layer, number of corneal endothelial cells and functional changes of the visual field Hypothesis: It is hypothesised that, based on its resolution and ease of use, SS-OCT is a suitable imaging technique to identify patients with or at risk of angle closure. It will be of value as an additional diagnostic instrument and may even replace gonioscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian race
2. 40-80 years
3. Willing and able to comply with scheduled visits and other study procedures
4. Signed informed consent
5. Participants derived from the study 'Caucasian patients with angle closure on SS-OCT' AND 1 or more of the following:

   * Irido-trabecular contact (ITC) in ≥2 quadrants as seen with SS-OCT in darkened conditions
   * Scleral spur angle (SSA) <20˚ (in 0 and 180º) AND anterior chamber depth (ACD) < 2.5 mm as seen with SS-OCT in darkened conditions
   * The fellow, non-treated eye in a patient after an acute primary angle closure (APAC) attack in the other eye. APAC is defined as an abrupt onset of symptomatic elevation of IOP resulting from total closure of the angle which is typically not self-limiting (although acute attacks can rarely resolve spontaneously).

Exclusion Criteria:

1. Any condition including (previous) intraocular laser/incisional surgery or medical procedure or treatment in ophthalmology
2. Any eye condition/abnormality that will affect the acquisition/reliability of measurement (results), (e.g. vitreous haemorrhage, uveitis, intraocular trauma, significant corneal opacity)
3. Unable to communicate properly or to understand instructions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will consist of Caucasian patients, aged 40-80 years. Patients will be recruited at the University Eye Clinic Maastricht, the Netherlands. All study participants are derived from the study 'Caucasian patients with angle closure on SS-OCT', METC 13-4-108.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Angle closure on gonioscopy | 3 weeks
  The percentage of subjects with angle closure on gonioscopy compared with angle closure on SS-OCT.

SECONDARY OUTCOMES:
intra-ocular pressure (IOP) | 3 weeks
  The secondary outcome measure is the percentage of patients with presence of an increased intra-ocular pressure (>21 mmHg) during the day or after dark provocation (IOP rise from baseline)

OTHER OUTCOMES:
Visual field loss | 3 weeks
  The percentage of patients with visual field loss on the HFA visual field.
Retinal nerve fiber layer thickness | 3 weeks
  The mean RNFL thickness will be measured.
Number of corneal endothelial cells | 3 weeks
  The mean number of corneal endothelial cells will be measured
Axial length | 3 weeks
  The mean axial length will be measured.
Anterior chamber angle parameters | 3 weeks
  Parameters analysed from SS-OCT images to determine the morphometric details of the anterior chamber will be measured and means will be calculated.
  For example AOD500, AOD750, TISA500, TISA750, ARA500, ARA750,TIA500, TIA750, ACD, LV

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Clinic Maastricht, Maastricht, Netherlands